CLINICAL TRIAL: NCT02155296
Title: Reducing Problem Behaviors Through PYD: An RCT of Restorative School Practices
Brief Title: RCT of the Restorative Practices Intervention
Acronym: RPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Joie Acosta, Behavioral Scientist, RAND
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1R01HD072235-01 (NIH); 1R01HD072235-01 (NIH)
Record Dates: First submitted 2014-05-29; First posted 2014-06-04 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Intervention Schools (Schools Receiving RPI); Control Schools (Schools Not Receiving RPI)
Keywords: positive youth development; restorative practices; school climate; social competency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Schools receiving RPI (Experimental): This arm contains schools receiving RPI. RPI offers a continuum of practices that range from informal (e.g., using affective statements that communicate feelings) to formal (e.g., hosting a restorative "circle" where participants are encouraged to express emotions and form emotional bonds). The "circles" or group meetings that are designed to take place between school staff and students, are the crux of RPI. School staff are encouraged to use the restorative practices to build relationships and resolve staff issues (restorative staff community), as well as when interacting with parents (restorative approach with families). All restorative practices encourage acting "with" youth and setting high expectations. When a school becomes proficient in all 11 essential practices it is officially recognized as a Restorative Practices School.
  Interventions: Behavioral: Restorative Practices Intervention
- Schools not receiving RPI (Experimental): This arm is the control arm and consists of schools that are not receiving RPI.
  Interventions: Behavioral: Restorative Practices Intervention

INTERVENTIONS:
Behavioral: Restorative Practices Intervention — RPI has the 3 core components of an optimal comprehensive positive youth development intervention:
  (1) sustained relationships with adults-RPI creates positive and sustained adult-youth relationships through teacher-student dialogue that occurs in "circles"; (2) skills building-RPI uses teachers and other school staff to coach students on 7 of the 11 essential practices; and (3) application of skills building-As students develop proficiency in the 7 essential practices they are coached to perform, school staff transfer responsibility for running the circles over to students. Restorative conferences for serious and or chronic behavior problems are the only circles that teachers continue to facilitate. Quasi-experimental studies have shown that schools implementing RPI have reductions in disciplinary referrals and school suspension.
  Other Names: Restorative Justice

SUMMARY:
The Restorative Practices Intervention (RPI), is a whole school environment intervention which is integrated into existing school practice (rather than 'added on') so does not compete with academic priorities; and it has some evidence supporting its effectiveness at improving school environment and promoting positive peer relationships. The specific aims of this investigator initiated study are to:

1. Assess the mechanisms of how RPI implementation influences the school environment;
2. Assess the effects of RPI on school staff perceptions of school climate and adolescents' reports of school connectedness, peer relationships, developmental outcomes (academic achievement and social competency) and problem behaviors (alcohol use, bullying, disciplinary referrals);
3. Assess the extent to which the positive effects of RPI on adolescents persist over time during the transition between middle and high school.

For the first time utilizing rigorous scientific methods, this study has the potential to document whether a whole-school intervention like RPI, that can be integrated into existing school practice, can affect both developmental outcomes and problem behaviors and whether the effects persist during the transition from middle to high school.

DETAILED DESCRIPTION:
Young adolescence is a critical time of development. Middle school youth (ages 11-14) experience biological, social, psychological, and cognitive changes and are exposed to a variety of risk factors that are mediated through their home and school environments and adult and peer relationships. It can be a time for positive growth and development, but also for both poor developmental outcomes (defined as limited social competency and poor academic achievement) and problem behaviors, including alcohol use, bullying, and school disciplinary referrals. Many programs that are delivered in schools, unfortunately, focus only on specific negative behaviors and deficits, like poor communication and decision making skills, and label adolescents as problems in need of fixing without leveraging the strengths and resiliency of youth. While many prevention programs can be effective at reducing or preventing negative behaviors-mostly in the short term-they do not tend to improve key developmental outcomes.This is in part because these programs are usually delivered as a stand-alone curriculum inserted into the school day and do not address the whole environment of a school. Also, these programs compete for time and resources with school priorities to meet academic standards. Transitions from elementary to middle and middle to high school, place adolescents at even greater risk for engaging in problem behaviors, underscoring the need for programs in the middle school years that promote positive developmental outcomes via programming that addresses the whole school environment.

Positive youth development (PYD) programs by contrast were developed to provide support, opportunities, and positive challenges for youth, to improve their developmental outcomes through leveraging youth's innate potential for positive growth and development (e.g., see articles). Comprehensive PYD programs (C-PYDs) address multiple dimensions shown to influence youth development (e.g., peers, school environment). Thus, these programs show promise in being able to mitigate negative behaviors like alcohol use and bullying, and promote developmental outcomes of social competency and academic achievement.

One C-PYD, the Restorative Practices Intervention (RPI), shows particular promise because it is a two-year, whole school environment intervention which is integrated into existing school practice (rather than 'added on') so does not compete with academic priorities; it is grounded in a strong theoretical basis (psychology of affect theory and ecological systems theory); and it has quasi-experimental evidence supporting its effectiveness at improving school environment and promoting positive peer relationships. Despite this evidence, questions remain about the exact mechanisms by which the results were achieved and whether results persist. Thus, more rigorous research is needed to assess RPI's impacts on academic achievement, social competencies, and problem behaviors; and the underlying program mechanisms that achieve positive outcomes across these areas. To improve the science of C-PYD evaluation, the goal for this 5-year study is to conduct a longitudinal randomized controlled trial of RPI in 16 schools to assess whether it impacts youth problem behaviors AND developmental outcomes. The study would be conducted under PA-08-241: Reducing Risk Behaviors by Promoting Positive Youth Development. The specific aims of this investigator initiated R01 are to:

1. Assess the mechanisms of how RPI implementation influences the school environment;
2. Assess the effects of RPI on school staff perceptions of school climate and adolescents' reports of school connectedness, peer relationships, developmental outcomes (academic achievement and social competency) and problem behaviors (alcohol use, bullying, disciplinary referrals);
3. Assess the extent to which the positive effects of RPI on adolescents persist over time during the transition between middle and high school.

For the first time utilizing rigorous scientific methods, this study has the potential to document whether a C-PYD like RPI, that can be integrated into existing school practice, can affect both developmental outcomes and problem behaviors and whether the effects persist during the transition from middle to high school. This information is critical as states are cutting funding to implement typical, stand-alone prevention programs and limiting the amount of time spent on non-academic prevention programs. This study will determine whether efficiencies can be gained by implementing C-PYD programs that have the potential to influence multiple outcome areas by influencing adolescents' developmental trajectory. As such, the study proposed here will impact the on-going debate about how to maximize federal/state resources devoted to middle school programming, and minimize the competition in-school prevention programs usually face with academic offerings. Findings also have the potential to advance the theory of PYD by empirically validating for the first time that restorative principles based on psychology of affect theory can be applied as an approach to promote PYD targeting a school environment.

ELIGIBILITY:
Inclusion Criteria:

* all students and staff in participating schools

Exclusion Criteria:

* anyone not in participating schools

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3516 (Actual)
Dates: Start 2014-08; Primary Completion 2019-01-12 (Actual); Study Completion 2019-01-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Perceptions of School Climate Post RPI and 1 year Post RPI | Baseline (pre-RPI), Post RPI, 1 year Post RPI (covers a time frame of 3 years total)
  This measure assesses teachers and students perceptions of: Consistency and Clarity of Rules and Expectations; Bullying; Teacher Support; and Student Input Into Decision Making. These dimensions can be aggregated into a single measure of school climate.
Change from Baseline in School Connectedness Post RPI and 1 year Post RPI | Baseline, Post RPI, 1 year Post RPI (covers a time frame of 3 years total)
  The school connectedness scale from the National Adolescent Health Study will be used to determine how close adolescents feel to their peers at this school, how happy they are to be at this school, whether they feel a part of the school, whether they feel teachers treat students fairly, and whether they feel safe at their school. The scale uses a five-point scale from "strongly agree" to "strongly disagree" to asses adolescents perception on 5 items and has shown strong internal consistency (alpha of 0.78).
Change from Baseline in Peer Relationships Post RPI and 1 year Post RPI | Baseline, Post RPI, 1 year Post RPI (covers a time frame of 3 years total)
  A scale developed by Acosta will be used to assess peer attachment and influence with nine items using a Likert rating of 1 (Never) to 6 (Always) measure how often their peers encouraged them to do well in school, how often they confide in peers, how often they would like to be the kind of person their peers are, how often they dress or act like their peers, and how often they consider how their peers will react before acting. Previous research has shown alphas of .71 for both subscales (attachment and influence) and sensitivity to detecting changes over time.
Change from Baseline in Social Competency Post RPI and 1 year Post RPI | Baseline, Post RPI, 1 year Post RPI (covers a time frame of 3 years total)
  The Social Skills Improvement System-Rating Scale (SSIS) will be used to assess students' perceptions of prosocial behavior in five domains: cooperation, assertion, responsibility, empathy, and self-control. The SSIS is a revision of the SSRS with updated national norms. Students self-rate their behavior on a 4-point frequency scale (0 = Never, 1 = Seldom, 2 = Often, and 3 = Almost Always). The SSIS-RS (for ages 13-18) was normed on a nationwide sample, all alpha coefficients are above 0.70, test-retest indices range from 0.77 to 0.92, and the SSIS is positively correlated with the SSRS (0.36).
Change from Baseline in Bullying Post RPI and 1 year Post RPI | Baseline, Post RPI, 1 year Post RPI (covers a time frame of 3 years total)
  The Communities That Care Survey questions will be used to assess prevalence of verbal, physical, and cyber bullying behaviors (perpetrator and victim). These questions were recently used in a study that found associations between bullying behaviors and alcohol use among middle school students. The scale assesses whether bullying behaviors that occurred in the past 30 days and the frequency of their occurrence (not at all, somewhat, and a whole lot).
Change from Baseline in Administrative Data Post RPI and 1 year Post RPI | Baseline, Post RPI, 1 year post RPI (covers a time frame of 3 years total)
  We will collect administrative data on academic achievement, and disciplinary referrals. These data will be collected through Maine's standardized school administrative data reporting system (Maine Educational Department Management System). Grades and incidences of detention, suspension, or expulsion will be used as indicators of academic achievement and disciplinary referrals, respectively. Standardized test scores were considered, but Maine has used a different test each cycle over the last few years, so data could not be used longitudinally. Further, our partners have confirmed that our schools do not grade on a distribution. Therefore, grades could improve school-wide as an outcome of RPI. Participating schools will also provide administrative data on students from the year before baseline, allowing us to have more information about student's prior trajectory of behavior.

SECONDARY OUTCOMES:
Dosage | Monthly during school year 1 and 2 (RPI Implementation)
  A Dosage Assessment completed by staff (on a monthly basis) will be used to track the frequency and duration of implementation of the 11 essential practices. For example, staff will be asked how often they used "I" statements over the past week or how long they spent in restorative circles over the past month.
Adherence | Monthly during school year 1 and 2 (RPI Implementation)
  Trainer Observations will be conducted at the 8 schools receiving RPI in-person on a monthly basis to assess adherence to the RPI implementation. Trainers will be observing RPI "circles", staff meetings, and parent-teacher nights to determine adherence to the 11 essential practices.
Participant Response | Once during school year 1 and once during school year 2 (RPI implementation)
  Implementation Surveys will measure participant response to RPI. Survey questions are designed to assess staff proficiency with each of 11 essential practices. For example, staff are asked to rate whether they can use affective statements in formal and informal interactions with students, and whether they can accurately assess whether their colleagues are using affective statements. RPI has used these measures extensively for quality improvement in previous studies and relies on these surveys to certify schools as a Restorative Practices school
Youth program quality assessment | Once during school year 1 and once during school year 2 (RPI implementation)
  The Youth Program Quality Assessment (YPQA) is an observational measure scored by an external rater that has 4 main scales: safe environment, supportive environment, interaction, and engagement-domains found to be critical to PYD interventions like RPI. A 2007 validation study found that across 32 rater pairs there was 78% perfect agreement at the item level, yielding an overall Kappa of .67, with alphas for subscales all over .69, indicating substantial overall agreement for items on this instrument. Validation studies also found that the YPQA had appropriate predictive validity needed to model process-outcome relationships where quality scores explain sizable amounts of variance in youth-level data.

CONTACTS AND LOCATIONS:
Overall Officials: Joie Acosta, Ph.D., Principal Investigator — RAND
Locations (13):
- United States (13):
  - Bath Middle School, Bath, Maine
  - Boothbay school, Boothbay Harbor, Maine
  - Bucksport school, Bucksport, Maine
  - Bonny Eagle school, Buxton, Maine
  - Ridge View school, Dexter, Maine
  - Molly Ockett, Fryeburg, Maine
  - Gorham school, Gorham, Maine
  - Jefferson Village school, Jefferson, Maine
  - Mt. Jefferson school, Lee, Maine
  - Maranacook school, Readfield, Maine
  - Oak Hill school, Sabattus, Maine
  - Skowhegan school, Skowhegan, Maine
  - Windham school, South Windham, Maine